CLINICAL TRIAL: NCT04104191
Title: The LIVMOR Data Collection Study for the Development and Validation of L-1000AF System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LIVMOR, Inc. (Industry)
Collaborators: Texas Health Dallas (Unknown); North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CIP-1001
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- L-1000AF System (Experimental): Software device on a wearable device used to detect irregular heart rhythms suggestive of Atrial Fibrillation
  Interventions: Device: L-1000AF System

INTERVENTIONS:
Device: L-1000AF System — The L-1000AF System is a wrist worn system that analyzes pulse rate data. The system identifies atrial fibrillation rhythms.

SUMMARY:
The LIVMOR Data Collection Study is a multicenter, IDE Exempt Study to generate a library of device-specific signals collected noninvasively. The study was not designed to evaluate specific hypothesis or endpoint, rather it was intended for data collection purposes to generate a library of raw clinical data that were retrospectively used for the development and subsequently the validation of the L-1000AF System. The L-1000AF System is a wrist worn system intended to provide continuous remote monitoring of atrial fibrillation (AF) episodes. The system is intended for use under the care of a physician and is not intended for the diagnosis of AF.

DETAILED DESCRIPTION:
LIVMOR is developing a series of wearable medical device systems intended to promote general wellness and help subjects and physicians manage various diseases that can benefit from increased visibility of physical activity, sleep, weight, blood pressure, stress/recovery levels and cardiac rhythms.

Data from human subjects is necessary to develop and validate LIVMOR devices. LIVMOR completed a multicenter, IDE Exempt Study to generate a library of device-specific signals collected non-invasively using components of the LIVMOR system and simultaneously acquired with ECG Holter data using a commercially available Holter monitor. Data from the analysis of the Holter monitor was adjudicated by physicians skilled in the analysis and interpretation of ECGs compared to the analysis from the LIVMOR AF Detection Algorithm to establish the sensitivity and specificity of the algorithm for detection of AF in comparison to ground truth.

The study was not designed to evaluate specific hypotheses or endpoint, rather it was intended for data collection purposes to generate a library of raw clinical data that were retrospectively used for the development and subsequently the validation of the L-1000AF System.

ELIGIBILITY:
Inclusion Criteria:

* Willing, able and sufficiently motivated to attend all study visits and participate in all study activities; and
* Physically and mentally capable of providing informed consent and are at least 18 years of age or of legal age to provide consent as required by local and national requirements.

Exclusion Criteria:

* Has any unstable or significant medical condition that is likely to interfere with study procedures or subjects medical care;
* Has any implantable electronic medical device;
* Has significant hearing, visual or cognitive impairment as determined by the Investigator; and
* Participating in any other clinical study without written consent from the Sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-14 (Actual)

PRIMARY OUTCOMES:
Concurrent Atrial Fibrillation | 10 minutes
  Simultaneous ECG monitoring indicating Atrial Fibrillation rhythm.
Detection of Atrial Fibrillation | 10 minutes
  A decision of Atrial Fibrillation detection in at least one 192-beat window.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Das, MD, Principal Investigator — Texas Health Dallas; Subhash Banerjee, MD, Principal Investigator — North Texas Veterans Healthcare System; Ken Persen, Study Director — LIVMOR, Inc.
Locations (2):
- United States (2):
  - VA North Texas Health Care System, Dallas, Texas
  - Texas Health Dallas, Dallas, Texas